CLINICAL TRIAL: NCT00120718
Title: The Effect of Fasudil on Vascular Function in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Mark A. Creager, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2002-P-000890
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Atherosclerosis; Hypercholesterolemia
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia | interventions — fasudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fasudil

SUMMARY:
The purpose of the study is to evaluate how the rho kinase inhibitor, fasudil, affects vascular function in patients with atherosclerosis and hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease
* Hyperlipidemia -OR-
* Healthy adults

Exclusion Criteria:

* Unstable angina, myocardial infarction or revascularization within 3 months
* Symptomatic heart failure
* Creatinine > 3.0 mg/dl
* Liver enzymes > 3X upper limit of normal
* Chronic hypoxia
* Significant anemia
* Chronic inflammatory disease
* Pregnancy
* Willing to withdraw statins for duration of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-06; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Vascular reactivity

SECONDARY OUTCOMES:
Rho kinase expression
Rho kinase activity
eNOS expression
eNOS activity
inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Creager, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States